CLINICAL TRIAL: NCT03734159
Title: Interest of Parasternal Block to Limit the Doses of Anesthetics Necessary for the Maintenance of Arterial Blood Pressure and Heart Rate in the Recommended Values During Sternotomy in Patients Undergoing Coronary Artery Bypass Graft
Brief Title: The Benefit of Local Anesthesia at the Sternum in Patients With Coronary Surgery
Acronym: PARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018/07
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2018-12

CONDITIONS: Coronary Bypass Graft Stenosis
Keywords: Regional Anesthesia; Sternotomy
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parasternal block (Experimental): preoperative parasternal block by ropivacaine injection
  Interventions: Drug: Ropivacaine
- physiological serum (Placebo Comparator): sodium chloride injection
  Interventions: Drug: sodium chloride 0.9%

INTERVENTIONS:
Drug: Ropivacaine — Injection of 60 ml of ropivacaine 0.25% divided into 4 injections of 15 ml (2 per side, between ribs 2 and 3 and between ribs 4 and 5)
  Arms: parasternal block
Drug: sodium chloride 0.9% — Injection of 60 ml of sodium chloride 0.9% divided into 4 injections of 15 ml (2 per side, between ribs 2 and 3 and between ribs 4 and 5)
  Arms: physiological serum

SUMMARY:
Patients undergoing coronary artery bypass grafting are at risk for perioperative myocardial ischemia. Episodes of tachycardia and hypertension, which are associated with an increase in myocardial oxygen consumption, are predictive events of these ischemia.

During cardiac surgery by sternotomy, some maneuvers, e.g. intubation, skin incision, sternotomy and cannulation, may be associated with tachycardia and/or increases in blood pressure despite an adequate level of anesthesia. Usually these episodes are controlled by the administration of a high-dose of anesthetic agents.

The parasternal block, by bolus or continuous infusion through a single catheter, showed its effectiveness on postoperative pain after sternotomy. It allows a blocking of anterior branches of intercostal nerves at the lateral edge of the sternum; branches in charge of innervation of the sternum and the overlying skin surface.

The preoperative parasternal block, once general anesthesia performed, could provide an effective level of locoregional anesthesia of the chest wall, thus limiting the occurrence of episodes of tachycardia and / or hypertension without having to resort to massive doses of anesthetic agents during sternotomy in patients undergoing coronary bypass surgery.

DETAILED DESCRIPTION:
This randomized double blinded placebo-controlled clinical trial will include patients undergoing coronary artery bypass grafting.

Locoregional anesthesia of the chest wall will be performed under ultrasound, once general anesthesia performed. A total volume of 60 ml of sodium chloride 0.9% (placebo group) or ropivacaine 0.25% (experimental group) divided into 4 injections of 15 ml (2 per side, between ribs 2 and 3 and between ribs 4 and 5) will be injected.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass graft requiring sternotomy other than re-interventions and combined surgeries
* Consent for participation
* Affiliation to the french social security system

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients under protection of the adults (guardianship, curator or safeguard of justice)
* Communication difficulties or neuropsychiatric disorder
* Neuropathic disease
* Constitutional coagulation disorders
* Kidney insufficiency
* Sensitivity to nonsteroidal anti-inflammatory drugs
* Hypersensitivity to local anaesthetics
* Chronic use of opioid analgesics
* Corticosteroid treatment or immunosuppressive therapy
* Autoimmune disease
* Chronic pain syndrome or fibromyalgia
* Emergency cardiac surgery
* Hypovolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Show that the preoperative realization of a parasternal block limites the posology of remifentanil administered during sternotomies to maintain blood pressure and heart rate within recommended ranges | Intraoperative period : from intubation to sternal retractor setup
  Maximal dose of remifentanil (morphine peak) required to maintain hemodynamic parameters (arterial blood pressure and heart rate) in the appropriate values during intubation, skin incision, sternotomy and sternal retractor setup

SECONDARY OUTCOMES:
Hemodynamic response : heart rate | Intraoperative period : from the start of general anesthesia maintenance to the fifth minute after sternal retractor setup
  Measure of heart rate in bpm
Hemodynamic response : arterial blood pressure | Intraoperative period : from the start of general anesthesia maintenance to the fifth minute after sternal retractor setup
  Measure of diastolic and systolic arterial blood pressure in mmHg
Hemodynamic response : patient state index | Intraoperative period : from the start of general anesthesia maintenance to the fifth minute after sternal retractor setup
  Measure of patient state index ranging from 0 to 100 (0=very deep anesthesia, 100=no hypnotic state)
Dose of hypnotic drug | Intraoperative period : from induction of anesthesia to skin closure
  Total amount of propofol administered during surgery
Dose of analgesic drug | Intraoperative period : from induction of anesthesia to skin closure
  Total amount of remifentanil administered during surgery
Inflammatory response | 7 days
  Serum concentrations of cytokines in pg/ml (composite : pro- (IL-6, IL-8, IL-1β, TNF-α, IFN-γ) and anti-inflammatory (IL-10) cytokines)
Pain level during extubation: Numeric scale | 8 hours
  Numeric scale of pain, ranging from 0 to 10 (0 = no pain, 10= worst possible pain)
Complications | 7 days
  Incidence of acute respiratory distress syndrome, pneumopathy, kidney failure or hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Bloc, MD, Principal Investigator — CMC Ambroise Paré
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bloc S, Perot BP, Gibert H, Law Koune JD, Burg Y, Leclerc D, Vuitton AS, De La Jonquiere C, Luka M, Waldmann T, Vistarini N, Aubert S, Menager MM, Merzoug M, Naudin C, Squara P. Efficacy of parasternal block to decrease intraoperative opioid use in coronary artery bypass surgery via sternotomy: a randomized controlled trial. Reg Anesth Pain Med. 2021 Aug;46(8):671-678. doi: 10.1136/rapm-2020-102207. Epub 2021 May 14. PMID 33990437